CLINICAL TRIAL: NCT00961883
Title: A Phase 1b Clinical Trial to Evaluate the Safety and Immunogenicity of Heterologous Prime/Boost Vaccine Regimens (NYVAC-B/rAd5 vs. rAd5/NYVAC-B) in Healthy, HIV-1 Uninfected, Ad5 Seronegative Adult Participants
Brief Title: Safety of and Immune Response to Prime/Boost Vaccine Regimens in Healthy, HIV-1 Uninfected, Ad5 Seronegative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); EuroVacc Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 078; 5U01AI068614 (NIH)
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; HIV Seronegativity; Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Thirty participants will receive injections in the following order: NYVAC-B for injections one and two, placebo for injection three, and rAd5 for the fourth and final injection. Two participants in this group will receive placebo vaccines only.
  Interventions: Biological: NYVAC-B; Biological: Placebo; Biological: rAd5
- 2 (Experimental): Fifteen participants will receive injections in the following order: rAd5 for injection one, placebo for injection two, and NYVAC-B for injections three and four. One participant in this group will receive placebo vaccines only.
  Interventions: Biological: NYVAC-B; Biological: Placebo; Biological: rAd5
- 3 (Experimental): Fifteen participants will receive injections in the following order: rAd5 for injection one, placebo for injection two, and NYVAC-B for injections three and four. One participant in this group will receive placebo vaccines only.
  Interventions: Biological: NYVAC-B; Biological: Placebo; Biological: rAd5
- 4 (Experimental): Fifteen participants will receive injections in the following order: rAd5 for injection one, placebo for injection two, and NYVAC-B for injections three and four. One participant in this group will receive placebo vaccines only.
  Interventions: Biological: NYVAC-B; Biological: Placebo; Biological: rAd5

INTERVENTIONS:
Biological: NYVAC-B — New York Vaccinia (NYVAC) vector for HIV-1, delivered intramuscularly by injection at a dose of 1 x 10 ^7 PFU
Biological: Placebo — Sodium Chloride for injection, delivered intramuscularly
Biological: rAd5 — Recombinant adenoviral serotype 5 (rAd5) vector vaccine, delivered by injection intramuscularly at a dose of 1 x 10^10 PFU
  Arms: 1; 4
Biological: rAd5 — Recombinant adenoviral serotype 5 (rAd5) vector vaccine, delivered by injection intramuscularly at a dose of 1 x 10^9 PFU
  Arms: 3
Biological: rAd5 — Recombinant adenoviral serotype 5 (rAd5) vector vaccine, delivered by injection intramuscularly at a dose of 1 x 10^8 PFU
  Arms: 2

SUMMARY:
Investigators will examine the safety of and immune responses to two vaccines expressing synthetic HIV proteins: NYVAC-B (a poxvirus), and rAd5 (an adenovirus). The study will compare responses in participants receiving NYVAC-B first, and rAd5 later, to those who receive rAd5 first, and NYVAC-B later. A different dose of rAd5 will be tested in each group.

DETAILED DESCRIPTION:
In order to halt the HIV pandemic an effective vaccine must be developed. In this study, investigators will examine the safety and immune response to a prime-boost strategy using two different vaccine regimens, NYVAC-B and rAd5.

Eighty participants will be recruited to this study. Participants will be randomly assigned to one of four different groups (study arms). Each group will receive both study vaccines and placebo but at different times. All NYVAC-B vaccine doses will be the same, but the doses of the rAD5 vaccine will differ from group to group. Some participants in each group will receive only placebo. Participants will visit the study clinic about 13 times over the course of 12 months and be contacted for follow-up for 4 years.

All study injections will be given in the same upper arm area. There will be a total of four injections during the course of the study. After each injection, participants will need to stay in the clinic for at least 25 minutes to check for any adverse reactions. Additionally, participants will need to monitor their own health on the evening after the injection and for the next three evenings, by taking their temperature and making notes of any noticed side effects. Tools will be provided to accomplish both of these tasks. During these few days following the injection, study investigators will need to maintain contact with participants (the participant will specify the best mode of contact).

Certain clinical procedures will be performed during the course of this study including regular HIV testing and counseling, physical exams, collection of blood and urine, pregnancy tests if applicable, questions about health and medications, questions about HIV risk and sexual behaviors, and any personal problems or benefits participants may have experienced from participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Assessment of understanding, including understanding of the Step Study results
* Willingness to receive HIV test results
* Amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by clinic staff as being "low risk" for HIV infection on the basis of sexual behaviors within the 12 months prior to enrollment. More information on this criterion is in the study protocol.
* Good general health
* Neutralizing antibody titers of Ad5 less than 1:18
* Hemoglobin count of 11.0 g/dL or more for female volunteers, and 13.0 g/dL or more for male volunteers
* White blood cell count of 3300 to 12000 cells/mm^3
* Total lymphocyte count of 800 cells/mm^3 or more
* Remaining differential either within institutional normal range or with site physician approval
* Platelets in the range of 125,000 to 550,000/mm^3
* Chemistry panel: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and creatinine values less than or equal to the institutional upper limits of normal
* HIV-uninfected
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine
* Not pregnant
* A volunteer who was born female must agree to consistently use effective contraception from at least 21 days prior to enrollment through the last protocol visit for sexual activity that could lead to pregnancy

Exclusion Criteria:

* Excessive alcohol use or chronic marijuana use, or any other illicit drug use within the 12 months prior to enrollment
* History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, within the 12 months prior to enrollment
* HIV vaccine received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, documentation of the identity of the study control/placebo must be provided to the HVTN 078 PSRT, who will determine eligibility on a case-by-case basis.
* Immunosuppressive medications received within 168 days before first vaccination
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 14 days after first injection
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 078 study
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion is in the study protocol.
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain
* Active syphilis infection
* Allergy to eggs and/or egg products
* History of, or known active cardiac disease
* Participants who have 2 or more specified cardiac risk factors as defined by the study. More information on this criterion is in the study protocol.
* ECG with clinically significant findings. More information on this criterion is in the study protocol.
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone
* Thyroidectomy, or thyroid disease
* Angioedema
* Hypertension
* Body mass index (BMI) equal to 40 and above or 35 and above with at least two of the following: systolic blood pressure greater than 140 mm Hg, diastolic blood pressure more than 90 mm Hg, current smoker, known hyperlipidemia
* Bleeding disorder
* Malignancy
* Seizure disorder
* Asplenia
* Psychiatric condition that precludes compliance with the protocol
* Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse events and serious adverse events meeting expedited adverse (EAE) criteria | Throughout study

SECONDARY OUTCOMES:
Magnitude and frequency of T-cell response as measured by ELISpot and/or intracellular cytokine staining (ICS) assay 2 weeks post 4th vaccination | At 2 Weeks following 4th Vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, Study Chair — CTU Lausanne; Pierre-Alexandre Bart, MD, Study Chair — Lausanne CRS
Locations (2):
- Switzerland (2):
  - BH10/513, Lausanne
  - BT06/614, Lausanne

REFERENCES:
- [Background] Gomez CE, Najera JL, Jimenez EP, Jimenez V, Wagner R, Graf M, Frachette MJ, Liljestrom P, Pantaleo G, Esteban M. Head-to-head comparison on the immunogenicity of two HIV/AIDS vaccine candidates based on the attenuated poxvirus strains MVA and NYVAC co-expressing in a single locus the HIV-1BX08 gp120 and HIV-1(IIIB) Gag-Pol-Nef proteins of clade B. Vaccine. 2007 Apr 12;25(15):2863-85. doi: 10.1016/j.vaccine.2006.09.090. Epub 2006 Oct 16. PMID 17113200
- [Background] Harari A, Bart PA, Stohr W, Tapia G, Garcia M, Medjitna-Rais E, Burnet S, Cellerai C, Erlwein O, Barber T, Moog C, Liljestrom P, Wagner R, Wolf H, Kraehenbuhl JP, Esteban M, Heeney J, Frachette MJ, Tartaglia J, McCormack S, Babiker A, Weber J, Pantaleo G. An HIV-1 clade C DNA prime, NYVAC boost vaccine regimen induces reliable, polyfunctional, and long-lasting T cell responses. J Exp Med. 2008 Jan 21;205(1):63-77. doi: 10.1084/jem.20071331. Epub 2008 Jan 14. PMID 18195071
- [Background] Liu J, O'Brien KL, Lynch DM, Simmons NL, La Porte A, Riggs AM, Abbink P, Coffey RT, Grandpre LE, Seaman MS, Landucci G, Forthal DN, Montefiori DC, Carville A, Mansfield KG, Havenga MJ, Pau MG, Goudsmit J, Barouch DH. Immune control of an SIV challenge by a T-cell-based vaccine in rhesus monkeys. Nature. 2009 Jan 1;457(7225):87-91. doi: 10.1038/nature07469. Epub 2008 Nov 9. PMID 18997770
- [Derived] Fischinger S, Cizmeci D, Deng D, Grant SP, Frahm N, McElrath J, Fuchs J, Bart PA, Pantaleo G, Keefer M, O Hahn W, Rouphael N, Churchyard G, Moodie Z, Donastorg Y, Streeck H, Alter G. Sequence and vector shapes vaccine induced antibody effector functions in HIV vaccine trials. PLoS Pathog. 2021 Nov 29;17(11):e1010016. doi: 10.1371/journal.ppat.1010016. eCollection 2021 Nov. PMID 34843602
- [Derived] Bart PA, Huang Y, Karuna ST, Chappuis S, Gaillard J, Kochar N, Shen X, Allen MA, Ding S, Hural J, Liao HX, Haynes BF, Graham BS, Gilbert PB, McElrath MJ, Montefiori DC, Tomaras GD, Pantaleo G, Frahm N. HIV-specific humoral responses benefit from stronger prime in phase Ib clinical trial. J Clin Invest. 2014 Nov;124(11):4843-56. doi: 10.1172/JCI75894. Epub 2014 Oct 1. PMID 25271627